CLINICAL TRIAL: NCT05513209
Title: Comparative Study Between Opioid Free Pterygopalatine Ganglion Block Based Multimodal Anesthesia Versus Conventional Opioid Based Multimodal Anesthesia for Tonsillectomy Operations
Brief Title: Opioid Free Pterygopalatine Ganglion Block Based Multimodal Anesthesia for Tonsillectomy Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00006379 TON
Record Dates: First submitted 2022-08-16; First posted 2022-08-24 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: PREVENTION OF POSTTONSILLECTOMY PAIN; DECREASE POSTTONSILLECTOMY NAUSEA AND VOMITTING; DECREASE POSTOPERATIVE HOSPITAL STAY

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid based multimodal anesthesia (Active Comparator): One hundred and twenty pediatric patients will do elective tonsillectomy or adenotonsillectomy surgery using opioid based multimodal anesthesia.
  Interventions: Procedure: opioid based multimodal anesthesia
- opioid free pterygopalatine ganglion block based multimodal anesthesia (Active Comparator): One hundred and twenty pediatric patients will do elective tonsillectomy or adenotonsillectomy surgery using opioid free pterygopalatine ganglion block based multimodal anesthesia.
  Interventions: Procedure: pterygopalatine ganglion block based multimodal anesthesia)

INTERVENTIONS:
Procedure: opioid based multimodal anesthesia — elective tonsillectomy or adenotonsillectomy surgery using opioid based multimodal anesthesia.
  Arms: opioid based multimodal anesthesia
Procedure: pterygopalatine ganglion block based multimodal anesthesia) — elective tonsillectomy or adenotonsillectomy surgery using opioid free pterygopalatine ganglion block based multimodal anesthesia.
  Arms: opioid free pterygopalatine ganglion block based multimodal anesthesia

SUMMARY:
intraoperative opioid administration versus intraoperative pterygopalatine ganglion block based opioid free anesthesia to compare outcomes such as postoperative administration of opioid rates of nausea and vomiting, Post Anesthesia Care Unit (PACU) length of stay

DETAILED DESCRIPTION:
Group A ;( opioid based multimodal anesthesia) One hundred and twenty pediatric patients will do elective tonsillectomy or adenotonsillectomy surgery using opioid based multimodal anesthesia.

Group B ;( opioid free pterygopalatine ganglion block based multimodal anesthesia) One hundred and twenty pediatric patients will do elective tonsillectomy or adenotonsillectomy surgery using opioid free pterygopalatine ganglion block based multimodal anesthesia.

For each patient, intraoperative hemodynamics, additional intraoperative analgesia required, the length of PACU stay, administration of postoperative opioids, administration of postoperative non-opioid analgesics, postoperative (visual analogue score) VAS score, will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 13 years old.
* Elective tonsillectomy or adenotonsillectomy surgery

Exclusion Criteria:

* Allergies to xylocaine.
* Developmental delays.
* Significant cognitive impairment.
* American Society of Anesthesiologists (ASA) Class 3 and 4.
* Patients who underwent any additional concurrent procedures such as lingual tonsillectomy.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
postoperative VAS score | EVERY HOUR AFTER SURGERY FOR 24 HOURS

SECONDARY OUTCOMES:
TOTAL AMOUNT OF OPIOD REQUIRED POSTOPERATIVELY | 24 HOURS AFTER SURGERY
INTRAOPERATIVE BLOOD PRESSURE | EVERY 10 MINUTES up to 1 hour
INTRAOPERATIVE HEART RATE | EVERY 10 MINUTES up to 1 hour
TOTAL AMOUNT OF GIVEN INTRAOPERATIVE OPIODS | DURING SURGERY
length of PACU stay | one day after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Ramymahrose, Cairo, Egypt